CLINICAL TRIAL: NCT00290732
Title: A Phase I Study Assessing the Feasibility and Safety of Intraductal Administration of Pegylated Liposomal Doxorubicin (Doxil) in Women With Breast Cancer
Brief Title: Liposomal Doxorubicin Before Mastectomy in Treating Women With Invasive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0503 CDR0000459502; P30CA006973 (NIH); JHOC-J0503 (Other: SKCCC at Johns Hopkins)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer; stage IV breast cancer; breast cancer in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraductal arm (Experimental): Participants received intraductal administration of dextrose or dextrose with pegylated liposomal doxorubicin hydrochloride (or PLD) prior to conventional surgery for breast cancer.
  Interventions: Drug: Intraductal arm
- Intravenous arm (Active Comparator): Participants receiving standard intravenous administration of pegylated liposomal doxorubicin prior to breast biopsy for drug concentrations.
  Interventions: Drug: Intravenous arm

INTERVENTIONS:
Drug: Intraductal arm — Patients will receive PLD intraductally according to the dose escalation schema (Dose Level -1=1 mg, Dose Level 1=2 mg, Dose Level 2= 5mg, Dose Level 3=10 mg). The PLD dose will be diluted in 5% dextrose in water and will be mixed for a total volume of 5 ml. The PLD will be administered via a breast duct (i.e., intraductally) using a microcatheter
  Other Names: Doxorubicin HCl Liposome Injection, Dox-SL, Doxil TM
  Arms: Intraductal arm
Drug: Intravenous arm — Blood samples and a breast tissue biopsy collected to look at levels of doxorubincol from patients receiving intravenous pegylated liposomal doxorubin to compare to the group receiving drug intraductally.
  Other Names: Doxorubicin HCl Liposome Injection, Dox-SL, Doxil TM
  Arms: Intravenous arm

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy in different ways, such as into the breast ducts, may kill more tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I trial is studying the side effects and best dose of liposomal doxorubicin when given before mastectomy in treating women with invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the feasibility, safety, and maximum tolerated dose of intraductal pegylated doxorubicin HCl liposome in women with invasive breast cancer awaiting mastectomy.

Secondary

* Determine the pharmacokinetics of intraductal pegylated doxorubicin HCl liposome, including serial plasma concentrations of doxorubicin and doxorubicinol and tissue concentrations in different portions of the breast at the time of surgery.

OUTLINE: This is a dose-escalation study.

Patients receive an intraductal injection of pegylated doxorubicin HCl liposome* on day 1. Patients undergo mastectomy 2-4 weeks later.

Cohorts of 3-6 patients receive escalating doses of pegylated doxorubicin HCl liposome* until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

NOTE: *The first cohort of 3 patients receive intraductal dextrose only followed by surgery as a feasibility study. An additional 3 patients receiving intravenous PLD will be enrolled in a pharmacokinetic control portion of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infiltrating carcinoma of the breast meeting any of the following criteria:

  * T1-3, any N disease
  * Proven ductal carcinoma in situ
* Unresected disease

  * Planned mastectomy as definitive surgical procedure

    * Known or suspected metastatic disease allowed provided mastectomy is planned
* Nonpalpable tumor allowed (e.g., initial T2-3 tumor that responded to preoperative therapy)
* No inflammatory breast cancer or other T4 features
* Successful baseline ductogram

  * Baseline nipple aspiration procedure must identify a duct productive of nipple aspirate fluid
  * No severe nipple retraction
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female patients
* Menopausal status not specified
* ECOG performance status 0-2
* Absolute neutrophil count ≥1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN
* AST and ALT ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant history of severe allergy to iodinated contrast material or debilitating anxiety that may not allow for a ductogram

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior preoperative chemotherapy, trastuzumab (Herceptin®), or hormonal therapy allowed provided it was completed 7-14 days prior to study treatment
* No prior radiation therapy, excisional biopsy, breast reduction, areolar surgery, or breast implant (present or past history of implant that was removed)
* No other prior procedure that may have altered the breast ductal system in the ipsilateral breast
* No other concurrent chemotherapy, radiotherapy, endocrine therapy, or biologic agents for breast cancer
* No other concurrent investigational drugs
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

REFERENCES:
- [Result] Stearns V, Mori T, Jacobs LK, Khouri NF, Gabrielson E, Yoshida T, Kominsky SL, Huso DL, Jeter S, Powers P, Tarpinian K, Brown RJ, Lange JR, Rudek MA, Zhang Z, Tsangaris TN, Sukumar S. Preclinical and clinical evaluation of intraductally administered agents in early breast cancer. Sci Transl Med. 2011 Oct 26;3(106):106ra108. doi: 10.1126/scitranslmed.3002368. PMID 22030751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2006 to October 2009, 19 women signed consent, and 17 women were enrolled in the intraductal portion of the study. An addition 3 women receiving standard intravenous PLD were enrolled in a pharmacokinetic contract portion.
Pre-assignment Details: Participants were not included after consent if eligibility criteria were not met (eg, lab values, performance status); an additional 2 subjects were consented but not included in the study population.
Groups:
- Intraductal Arm- 0 mg PLD: Participants received intraductal administration of dextrose prior to conventional surgery for breast cancer.
- Intraductal Arm- 2 mg PLD: Participants received intraductal administration of pegylated liposomal doxorubicin hydrochloride (or PLD), 2 mg, prior to conventional surgery for breast cancer.
- Intraductal Arm- 5 mg PLD: Participants received intraductal administration of pegylated liposomal doxorubicin hydrochloride (or PLD), 5 mg, prior to conventional surgery for breast cancer.
- Intraductal Arm- 10 mg PLD: Participants received intraductal administration of pegylated liposomal doxorubicin hydrochloride (or PLD), 10 mg, prior to conventional surgery for breast cancer.
Period: Overall Study
Arm/Group | Intraductal Arm- 0 mg PLD | Intraductal Arm- 2 mg PLD | Intraductal Arm- 5 mg PLD | Intraductal Arm- 10 mg PLD | Intravenous Arm
Started | 3 | 4 | 4 | 6 | 3
Completed | 3 | 3 | 3 | 6 | 3
Not Completed | 0 | 1 | 1 | 0 | 0
Not completed — Inability to instill drug intraductally. | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraductal Arm | Intravenous Arm | Total
Number analyzed (Participants) | 17 | 3 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 3 | 18
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 3 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Maximum tolerated dose (MTD) of administering pegylated liposomal doxorubicin (PLD) into one duct of women with breast cancer awaiting mastectomy. MTD reflects highest dose of drug that did not cause Dose Limiting Toxicity (DLT) in more than 30% of patients.
Time Frame: Until up to 30 days after PLD administration
Population: Participants received intraductal administration of dextrose prior to conventional surgery for breast cancer.
Measure: Number; unit: milligrams
Arm/Group | Intraductal Arm
Number analyzed (Participants) | 15
milligrams | 10

2. Secondary Outcome: Concentrations of Doxorubicin in Blood (Plasma) at Definitive Surgery
Description: Due to the limited number of samples and detectable levels, the maximum concentration of doxorubicin in blood (plasma) across all the participants in each group is reported.
Time Frame: Baseline, 4 hrs, day2/24 hrs, day 8, day of surgery/biopsy
Population: Participants in whom blood and/or tissue samples were collected at surgery or breast biopsy.
Measure: Number; unit: nM
Groups:
- Intraductal Arm- 2 mg PLD: Participants received intraductal administration of dextrose with pegylated liposomal doxorubicin hydrochloride (or PLD), 2 mg, prior to conventional surgery for breast cancer.
- Intraductal Arm- 5 mg PLD: Participants received intraductal administration of dextrose with pegylated liposomal doxorubicin hydrochloride (or PLD), 5 mg, prior to conventional surgery for breast cancer.
- Intraductal Arm- 10 mg PLD: Participants received intraductal administration of dextrose with pegylated liposomal doxorubicin hydrochloride (or PLD), 10 mg, prior to conventional surgery for breast cancer.
Arm/Group | Intraductal Arm- 0 mg PLD | Intraductal Arm- 2 mg PLD | Intraductal Arm- 5 mg PLD | Intraductal Arm- 10 mg PLD | Intravenous Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3
nM
  Doxorubicin, max | 0 [0 to 0] | 28.5 | 18.3 | 902.0 | 79300
  Doxorubicinol, max | 0 | 0 | 0 | 36.9 | 8090

3. Secondary Outcome: Concentrations of Doxorubicin in Tissue at Definitive Surgery
Description: Due to the limited number of samples and detectable levels, the maximum concentration of doxorubicin in tissue across all the participants in each group is reported.
Time Frame: Day of surgery/biopsy
Population: Participants in whom blood and/or tissue samples were collected at surgery or breast biopsy.
Measure: Number; unit: nmol/g
Arm/Group | Intraductal Arm- 0 mg PLD | Intraductal Arm- 2 mg PLD | Intraductal Arm- 5 mg PLD | Intraductal Arm- 10 mg PLD | Intravenous Arm
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3
nmol/g
  Doxorubicin, max | 0 | 0 | 1.73 | 10.82 | 0.21
  Doxorubicinol, max | 0 | 0 | 0.09 | 5.26 | 0

ADVERSE EVENTS:
Time Frame: After definitive surgery
Description: Note: Adverse events were not collected in the intravenous group/arm; only the concentration of doxorubicin in tissue applied to this group of participants.
Groups:
- Intravenous Arm: Note: Adverse events were not collected in the intravenous group/arm; only the concentration of doxorubicin in tissue applied to this group of participants.
Arm/Group | Intraductal Arm- 0 mg PLD | Intraductal Arm- 2 mg PLD | Intraductal Arm- 5 mg PLD | Intraductal Arm- 10 mg PLD | Intravenous Arm
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/6 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraductal Arm- 0 mg PLD (N=3) | Intraductal Arm- 2 mg PLD (N=3) | Intraductal Arm- 5 mg PLD (N=3) | Intraductal Arm- 10 mg PLD (N=6) | Intravenous Arm (N=0)
Dermatology other (right areolar eschar) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Eschar/necrosis in the region of the remaining areola of the right breast post-mastectomy.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intraductal Arm- 0 mg PLD (N=3) | Intraductal Arm- 2 mg PLD (N=3) | Intraductal Arm- 5 mg PLD (N=3) | Intraductal Arm- 10 mg PLD (N=6) | Intravenous Arm (N=0)
Breast fullness (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Breast or nipple pain/discomfort (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 3 (3) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
Duct cannulation was not successful in all participants; possibly due to extensive disease or prior excisional biopsy (2 subjects).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No